CLINICAL TRIAL: NCT03526159
Title: A Pilot Study of the Restoration of Functional Laminin 332 in JEB Patients With Nonsense Mutations After Topical and Intravenous Gentamicin Treatment
Brief Title: Gentamicin for Junctional Epidermolysis Bullosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, David Woodley, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-18-00290
Record Dates: First submitted 2018-04-17; First posted 2018-05-16 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Junctional Epidermolysis Bullosa
Keywords: Herlitz; Laminin 332; Laminin beta 3; JEB
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gentamicin Sulfate (Experimental): IV Arm:
  7.5 mg/kg gentamicin once daily for 14 days.
  Topical Arm:
  0.5% gentamicin ointment applied twice daily for 14 days to selected skin sites.
  Interventions: Drug: Gentamicin Sulfate

INTERVENTIONS:
Drug: Gentamicin Sulfate — Gentamicin (formulated as gentamicin sulfate) is a well-known, well-characterized antibiotic that has been used for four decades as a treatment against gram negative bacteria. It, like other aminoglycoside antibiotics, has the well documented added potential to facilitate readthrough of premature termination codons in eukaryotic cells and organisms.
  Other Names: Gentamicin

SUMMARY:
Herlitz junctional epidermolysis bullosa (H-JEB), an incurable, fatal, inherited skin disease, is caused by loss-of-function mutations in the LAMA3, LAMB3 or LAMC2 genes, resulting in loss of laminin 332 and poor epidermal-dermal adherence. Eighty percent of H-JEB patients have LAMB3 mutations and about 95% of these are nonsense mutations. The investigators recently demonstrated that gentamicin readily induced nonsense mutation readthrough and produced full-length laminin beta3 in several nonsense mutations tested. Importantly, the gentamicin-induced laminin beta3 restored laminin 332 assembly, secretion, and deposition into the dermal-epidermal junction (DEJ). Newly induced laminin 332 reversed abnormal H-JEB cellular phenotypes. Herein, the investigators propose the first clinical trial of gentamicin (by topical and intravenous administration) in JEB patients with nonsense mutations. The milestones will include restored laminin 332 and hemidesmosomes at the DEJ, improved wound closure, and the absence of significant gentamicin side effects.

DETAILED DESCRIPTION:
Three subjects (adults and children of any age) will receive topical gentamicin to be applied to select skin sites.

Three subjects (adults and children of any age) will receive intravenous (IV) gentamicin infusions.

Patients will be assessed for Primary and Secondary endpoints during follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. JEB patients with nonsense mutations in the LAMB3 gene in either one or two alleles.

Exclusion Criteria:

1. JEB patients who do not have nonsense mutations in the LAMB3 gene in either allele.
2. Pre-existing known auditory impairment.
3. Pre-existing known renal impairment.
4. Pre-existing known allergies to aminoglycosides or sulfate compounds.
5. Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Increased laminin beta 3 / laminin 332 expression as assessed by immunofluorescence. | 3 months
  New or increased staining of the target protein, laminin 332, in sections of skin biopsies obtained during follow-up visits in comparison with baseline biopsies. Five micron cryosections will be probed with three different antibodies against laminin 332. Patient samples along with normal control samples will be compared. Mean fluorescence intensity will be calculated for each sample and antibody using ImageJ software. Percent expression relative to normal human skin (set to 100%) will be calculated for each patient sample. Any statistically significant increase in (p value < 0.05) over baseline will be considered improvement.
Incidence of Treatment-Emergent Adverse Events | 3 months
  The total number of adverse events and serious adverse events will be recorded and enumerated for each study participant. Gentamicin in high doses is associated with ototoxicity and nephrotoxicity. Audiometry and creatinine clearance tests will be performed throughout the study to monitor for the emergence of any treatment-related adverse events. In addition, as this treatment may result in the production of a protein that is hasn't been present in the patient's system, commercial ELISA tests will be performed on serum samples to test for the emergence of circulating anti-laminin 332 antibodies. Adverse events include a decline of >15 dB on pure tone audiometry at 2 consecutive frequencies, creatinine clearance <60ml/min, presence of antibodies to laminin 332, and for IV gentamicin recipients, serum gentamicin peak levels above 40 ug/ml and trough levels above 2 ug/ml.
Generation of new hemidesmosomes as assessed by electron microscopy. | 3 months
  Any new hemidesmosomes detected by electron microscopy in post-treatment skin biopsies will be enumerated and compared to baseline.

SECONDARY OUTCOMES:
Improved wound closure. | 3 months
  Participants in the Topical arm will treat and monitor specific test sites, along with untreated control sites, selected during their baseline visits. Photographs will be used to assess the size of open erosions. Wound areas (treated and untreated) (cm2) will be measured using computer-assisted planimetry of digital photographs taken throughout the study.
Reduction in blistering | 3 months
  Participants in the Topical arm will treat and monitor specific test sites, along with untreated control sites, selected during their baseline visits. Photographs and patient diaries will be used to assess the number of blisters that appear at the test sites as well as whether the wound had closed during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Mosallaei D, Hao M, Antaya RJ, Levian B, Kwong A, Cogan J, Hamilton C, Schwieger-Briel A, Tan C, Tang X, Woodley DT, Chen M. Molecular and Clinical Outcomes After Intravenous Gentamicin Treatment for Patients With Junctional Epidermolysis Bullosa Caused by Nonsense Variants. JAMA Dermatol. 2022 Apr 1;158(4):366-374. doi: 10.1001/jamadermatol.2021.5992. PMID 35234826